CLINICAL TRIAL: NCT06863974
Title: High-throughput Omic Technology for Identification of Biomarkers of Relapsing Acute Disseminated Encephalomyelitis in the Immune Cell Network
Brief Title: High-throughput Omic Technology for Identification of Biomarkers of Relapsing Acute Disseminated Encephalomyelitis in Immune Cell Network
Acronym: HOT-BRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A02732-45
Record Dates: First submitted 2024-12-16; First posted 2025-03-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Disseminated Encephalomyelitis; Encephalitis Autoimmune
MeSH Terms: conditions — Encephalomyelitis, Acute Disseminated; Autoimmune Diseases of the Nervous System | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Prospective recruitment requires pre-inclusion because the characterization of antibodies allowing patients to be classified into these 3 groups is only done at a later stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADEM non-MOGAD (Experimental): Non-MOGAD ADEM control group of 5 patients with anti-MOG antibody-negative ADEM
  Interventions: Other: Blood test
- ADEM MOGAD (Active Comparator): Single-phase and multi-phase ADEM MOGAD units respectively
  Interventions: Other: Blood test
- MOGAD non-ADEM (Experimental): MOGAD non-ADEM central nervous system demyelinating neuroinflammatory control group (anti-MOG antibody-positive optic neuritis or myelitis) of 5 patients
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Drawing blood to realize biomarkers of disease course of MOGAD-ADEM and pathophysiology of ADEM (and MOGAD) : cellular and molecular signatures, inflammatory signaling.

SUMMARY:
Acute disseminated encephalomyelitis (ADEM) is a neuroinflammatory disorder of the central nervous system, manifesting itself as impaired consciousness, even to the point of coma, and multifocal neurological deficits. ADEM is the most common encephalitis in children. Moreover, 50-65% of ADEM in children is associated with the presence of anti-MOG antibodies (MOGAD). In fact, ADEM is the most frequent clinical presentation of MOGAD in children, 50-75% before the age of 10. The risk of recurrence is higher in pediatric MOGAD of ADEM manifestation, up to 30%, compared to myelitis or optic neuritis. Multiphasic MOGAD are more frequently associated with sequelae in 50-69% of cases, versus 4-32% for monophasic forms. In ADEM, cognitive and epileptic sequelae predominate. The 2020 European consortium and the 2022 national diagnosis and care protocol recommend the introduction of disease-modifying therapies as early as the second attack of the disease, or in the event of distant sequelae, in order to limit relapses and sequelae. However, these treatments take several months to take effect.

There is currently no reliable predictive factor for MOGAD recurrence other than the persistence of an elevated blood anti-MOG antibody level (≥1:1280) at 1 year. The aim of this study is therefore to identify biomarkers associated with MOGAD recurrence from the first attack. To this end, we will study the transcriptome of circulating blood mononuclear cells by single-cell next-generation RNA sequencing in children with anti-MOGAD neuroinflammatory relapses. Anticipating the multiphasic trajectory of the disease would enable the introduction of early disease-modifying therapy to prevent recurrences and long-term sequelae. Furthermore, the discovery of a molecular and/or cellular signature would provide a better understanding of the pathophysiology of ADEM and MOGAD.

ELIGIBILITY:
Inclusion criteria:

Prospective recruitment Pre-inclusion criteria

* Age at inclusion between 1 and 18 years (included)
* First demyelinating event at inclusion, such as ADEM encephalitis, optic neuritis (NORB) or myelitis, or a combination of these conditions.
* Informed consent signed by patient's legal representative
* Patient affiliated to or benefiting from a social security scheme Inclusion criteria (confirmation of inclusion and follow-up in one of 3 groups)
* MOGAD/ADEM group: presence of serum anti-MOG antibodies and diagnosis of ADEM (according to the International Pediatric Multiple Sclerosis Society Group (IPMSSG) criteria revised in 2013) at the first demyelinating attack.
* Non-MOGAD/ADEM group: anti-MOG antibodies negative and diagnosis of ADEM at first demyelinating attack.
* MOGAD/non-ADEM group: presence of serum anti-MOG antibodies and diagnosis of myelitis and/or NORB at first demyelinating attack.

Retrospective recruitment General inclusion criteria

* Age at inclusion between 1 and 18 years (inclusive)
* Inclusion (signed consent of the patient's legal representative) in the biocollection from which the samples were taken at the latest at the time of management of a first demyelinating event of the ADEM encephalitis, optic neuritis (NORB) or myelitis type, or a combination of these disorders.
* PBMC collected at the time of the first demyelinating event before any immunomodulatory treatment, cryopreserved and available in the biocollection.
* Depending on the date of inclusion (if inclusion beyond 6 to 24 months after the first demyelinating event), samples taken at 6 months and then 24 months after the first demyelinating event available in the biocollection for the analyses planned in the study.
* Informed consent signed by patient's legal representative
* Patient affiliated to or benefiting from a social security scheme

Inclusion criteria specific to the 3 study groups

* MOGAD/ADEM group: presence of serum anti-MOG antibodies and diagnosis of ADEM (according to the International Pediatric Multiple Sclerosis Society Group (IPMSSG) criteria revised in 2013) at the first demyelinating attack.
* Non-MOGAD/ADEM group: anti-MOG antibodies negative and diagnosis of ADEM at first demyelinating attack.
* MOGAD/non-ADEM group: presence of serum anti-MOG antibodies and diagnosis of myelitis and/or NORB at first demyelinating attack.

Non-inclusion criteria (prospective or retrospective recruitment):

* Immunosuppressive therapy in the 6 months prior to treatment for a first demyelinating event.
* Systemic corticosteroid therapy or immunomodulating doses of IV polyvalent immunoglobulin or plasma exchange within 3 months prior to treatment for a first demyelinating event.
* Brain MRI not performed at diagnosis of first demyelinating event
* Poor understanding of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-16 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood sample | Inclusion, 6 months, 24 months
  1 tube (approx. 5 mL) for children under 12 kg, 2 tubes (approx. 10 mL) for children between 12 kg and 20 kg, 4 tubes (approx. 20 mL) for children over 20 kg.
  Collected tubes are transferred to the investigator's Biological Resource Center (BRC) for sample preparation of the biocollection, if accepted in the consent form, and preparation of circulating blood mononuclear cells (PBMC).
Age | Inclusion
Personal or family history of inflammatory or dysimmune disease | Inclusion
Weight | Inclusion, 6 months, 24 months
  Weight (kg)
EDSS (Expanded Disability Status Scale) | Inclusion, 6 months, 24 months
  The neurological examination is divided into eight functional systems, 4 major (pyramidal, cerebellar, sensory, brainstem), 4 minor (sphincter, vision, mental and other).
  A numerical score of increasing severity (0 to 6 or 7) is given to each functional system (FS). The overall scale score is measured on a 20-level scale (0 to 10 per half-point). Up to level 3.5, the score obtained in each FS (Functional System) and the number of FS reached automatically determine the EDSS score. From 4 to 7, the definition of each level is also given by the walking disability (ability to walk without stopping, need for assistance).
Neurological episodes consistent with demyelinating relapse since previous visit | 6 months, 24 months
  Number, date, neurological symptoms including chronic fatigue unusual for an individual of the same age, diagnosis of demyelinating relapse, type, hospitalization, treatment with intravenous corticosteroid bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Nail Benallegue, MD, Principal Investigator — University Hospital, Angers
Locations (6):
- France (6):
  - CHU d'Angers, Angers
  - Univesity Hostipal of Brest, Brest
  - Univesity Hostipal of APHP, Le Kremlin-Bicêtre
  - Univesity Hostipal of Nantes, Nantes
  - Univesity Hostipal of Rennes, Rennes
  - Univesity Hostipal of Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).